CLINICAL TRIAL: NCT06068244
Title: 3D-Printed Crowns Versus Prefabricated Zirconia Crowns for the Restoration of Pulpally-treated Primary Molars; Randomized Clinical Trial and In-Vitro Study
Brief Title: 3D-printed Crowns Versus Zirconia Crowns for Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esaad El Nagar, Assistant lecturer at pediatric dentistry and dental public health department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED23-1D
Record Dates: First submitted 2023-09-08; First posted 2023-10-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries in Children
Keywords: "zirconia crowns"; "pulpotomy"; "3 dimension printed crowns"

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed crowns (Experimental): Participants received 3D printed resin crowns
  Interventions: Other: 3D printed crowns
- Zirconia crowns (Active Comparator): Participants received ready made zirconia crowns
  Interventions: Other: Zirconia crowns

INTERVENTIONS:
Other: 3D printed crowns — 3D printed crowns
  Arms: 3D printed crowns
Other: Zirconia crowns — Nu smile zirconia crowns
  Arms: Zirconia crowns

SUMMARY:
The aim of the present study is to compare between 3D-printed crowns and prefabricated zirconia crowns for restoring pulpally-treated primary molars regarding the following aspects:

1. In vivo:

   Evaluate the clinical outcome of 3D printed crowns in comparison to prefabricated zirconia crowns in pulpally-treated primary molars as well as parent satisfaction.
2. In vitro:

Comparative analysis of fracture resistance and marginal gap of 3D printed crowns and prefabricated zirconia crowns

DETAILED DESCRIPTION:
in vitro part :

All selected primary molars should fulfill the following criteria:

1. Freshly extracted molars with at least three sound walls.
2. Retain at least one third of their roots Teeth preparation All soft tissue debris will be removed with a hand scaler and teeth will be disinfected, and then stored in distilled water at 4 degrees Celsius until the start of the study.

Pulpotomy procedures will be performed to the extracted molars and the molars will be filled. Then, they will be randomly allocated into two groups.

Group 1: Will receive 3D-printed crowns Group 2: Will receive prefabricated zirconia crowns The specimens will be embedded perpendicularly in Polyvinyl chloride (PVC) cubes with the occlusal surface parallel to the ground using acrylic resin extending 2mm below the cementoenamel junction.

Evaluations: teeth in both groups will be evaluated for the following:

1. Marginal gap:

   Precementation measurements of the cervical vertical marginal discrepancies will be performed before cementation., Four optical images for each specimen will be captured using a stereomicroscope (Wild 400, Switzerland) at a 32× magnification. Images will then be transferred to the computer software for image analysis.
2. Fracture Resistance:

An axial loading condition through the functional cusp will be defined in the mechanical failure description. Failure-to-fracture strength will be tested with a universal testing machine (LLOYD machine) at a 0.5 mm/sec crosshead speed. Application of a round-end vertical loading tip on the occlusal third of a specimen fixed into a loading apparatus as functional loading simulation.

in vivo part : Teeth will be polished using a polishing paste and brush, and dried before being examined.

A dental mirror will be used for clinical examination under light emitting diode (LED) illumination to confirm the fulfillment of the inclusion criteria of the patient's selection.

* The molars will be randomly allocated into two equal treatment groups 23/each):

  1. Group 1: 3D-printed crowns
  2. Group 2: prefabricated zirconia crowns

     Pulpotomy procedure for both groups:

  <!-- -->

  1. Local anesthesia will be administered.
  2. Teeth will undergo pulpotomy procedure' as follows:
* Caries removal will be done using a large size 4 round bur, mounted onto a high-speed hand piece with constant coolant.
* All access cavity walls will be flared to allow complete exposure of the pulp chamber, and easy undisturbed access to the canals, followed by removal of all the soft pulpal tissue tags by a sharp spoon shaped excavator.
* Bleeding control will be done using moist cotton pellet with gentle pressure.
* Formocresol will be applied using a cotton pellet for 3-5 mins, for fixation.
* The pulp chamber will be filled with re-inforced zinc oxide and eugenol that will be mixed according to manufacturer's instructions.
* Analgesics will be prescribed to the patient to be taken when needed.

Intervention Group 1:

1. Crown reduction: The teeth will be prepared using taper diamond bur with round end for buccal, lingual, mesial, and distal wall for 0.8- 1 mm, producing a chamfer margin circumferentially, and then, reduction of the occlusal surface will be done using a round wheel to produce occlusal clearance of 1.5 mm.
2. Impression for the preparation will be taken using putty and light poly vinyl siloxane material.
3. The impression will be sent to the lab and the patient will be dismissed.
4. The preparation will be optically scanned in the lab and the crown will be digitally designed using computer designing software.
5. The crown will be printed using 3D printer.
6. The 3D printed crown will be cemented in the 2nd visit.

Control: Group 2:

1. Crown reduction:

   * In order to compensate for the thickness of zirconia crown, reduction will be performed on the mesial, distal, buccal and lingual surfaces of the tooth for 0.7-1.75mm. Reduction will be performed using fine needle stone in the beginning to free the contact from the adjacent teeth then followed by reduction of the other surfaces using a diamond stone.
   * Reduction of the occlusal surface will be performed using a flame stone or wheel stone to produce occlusal clearance of 1.5- 2 mm.
   * All line angles will be checked to remove any sharp line angles.
2. Selection of the matching size from zirconia crowns will be made taking into consideration that the preparation must be free from any undercuts to avoid crown fracture.
3. After checking the selected size of the crowns, it will be removed, dried and cemented to the tooth using resin cement.

Method of evaluation:

After cementation , at baseline ,3rd ,6th and 12th months evaluation of the crowns will be performed clinically using the modified U.S. Public Health Service criteria for retention, marginal integrity and gingival health for both groups. Also, parental satisfaction will be evaluated at end of the study using 5-point likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the study should stratify to the following criteria:

  * Age range of children from 4 -7 years.
  * Having at least one vital primary molar with deep carious lesion indicated for pulpotomy or pulpectomy.
  * The expected exfoliation date of the selected primary teeth must be more than 12 months from the start date of the study.

Exclusion Criteria:

* a) Uncooperative children who needs sedation or general anesthesia. b) Children with physical, intellectual disability or medical conditions that may complicate treatment.

  c) Teeth with poor prognosis due to the presence of an abscess or a sinus, mobility or advanced bone resorption.

  d) Presence of internal or external root resorption.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Gingival health (gingival index) | 1 year follow up for vivo part only
  Gingival index and plaque index
  A gingival index, based on the Loe and Silness scoring criteria (1963). It will be measured by gently inserting the tip of a periodontal probe into the sulcus surrounding each tooth. Scoring as followed:
  0 = Normal (Absence of inflammation)
  1. = Mild gingivitis (slight change in color, slight edema. No bleeding on probing)
  2. = Moderate gingivitis (redness, edema and glazing. Bleeding on probing)
  3. = Severe gingivitis (marked redness and edema; ulceration; tendency to spontaneous bleeding)
     * Gingival index and plaque index.
plaque index | 1year follow up
  Plaque index (PI) (Silness and Loe) PI 0: No observable plaque PI 1: A thin film of plaque is detected at the gingival margin by running a probe or explorer across the tooth surfaces PI 2: A moderate amount of plaque is detected along the gingival margin. Plaque is visible clinically.
  PI 3: Heavy plaque accumulation is detected at the gingival margin and in the interdental Plaque index (PI) (Silness and Loe) PI 0: No observable plaque PI 1: A thin film of plaque is detected at the gingival margin by running a probe or explorer across the tooth surfaces PI 2: A moderate amount of plaque is detected along the gingival margin. Plaque is visible clinically.
  PI 3: Heavy plaque accumulation is detected at the gingival margin and in the interdental
Marginal integrity | 1yeat follow up
  by visual inspection and explorer Alfa: Explorer does not catch or has one way catch when drawn across the restoration/tooth interface.
  Bravo: Explorer falls into crevice when drawn across the restoration/tooth interface, Dentin is not exposed; clinically acceptable.
  Charlie: Dentin or base is exposed along the margin; clinically unacceptable.
crown retention | one year follow up
  Alpha: Bonded Bravo: Debonded Charlie: Lost
In vitro marginal gap | Immediately after samples preparation
  micrometers
in vitro fracture resistance | Immediately after samples preparation
  newton

SECONDARY OUTCOMES:
parent satisfaction | immediately after cementation of crowns
  5-point likert scale.1-very dissatisfied; 2-dissatisfied; 3-neutrally satisfied; 4-satisfied; 5-very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Geham Gaber allam, Study Director — Assistant professor
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamrah MH, Mokhtari S, Hosseini Z, Khosrozadeh M, Hosseini S, Ghafary ES, Hamrah MH, Narges Tavana. Evaluation of the Clinical, Child, and Parental Satisfaction with Zirconia Crowns in Maxillary Primary Incisors: A Systematic Review. Int J Dent. 2021 Jul 5;2021:7877728. doi: 10.1155/2021/7877728. eCollection 2021. PMID 34285695
- [Background] Al-Halabi MN, Bshara N, Nassar JA, Comisi JC, Rizk CK. Clinical Performance of Two Types of Primary Molar Indirect Crowns Fabricated by 3D Printer and CAD/CAM for Rehabilitation of Large Carious Primary Molars. Eur J Dent. 2021 Jul;15(3):463-468. doi: 10.1055/s-0040-1721905. Epub 2021 Feb 3. PMID 33535245
- [Background] Abuelniel G, Eltawil S. Clinical and Radiographic Evaluation of Stainless Steel versus Zirconia Crowns on Primary Molars: Randomized Controlled Trial. Egypt Dent J. 2018;64(2):977-89.
- [Background] Mathew MG, Roopa KB, Soni AJ, Khan MM, Kauser A. Evaluation of Clinical Success, Parental and Child Satisfaction of Stainless Steel Crowns and Zirconia Crowns in Primary Molars. J Family Med Prim Care. 2020 Mar 26;9(3):1418-1423. doi: 10.4103/jfmpc.jfmpc_1006_19. eCollection 2020 Mar. PMID 32509626
- [Background] Ludwig KH, Fontana M, Vinson LA, Platt JA, Dean JA. The success of stainless steel crowns placed with the Hall technique: a retrospective study. J Am Dent Assoc. 2014 Dec;145(12):1248-53. doi: 10.14219/jada.2014.89. PMID 25429038
- [Background] Attari N, Roberts JF. Restoration of primary teeth with crowns: a systematic review of the literature. Eur Arch Paediatr Dent. 2006 Jun;7(2):58-62; discussion 63. doi: 10.1007/BF03320816. PMID 17140529
- [Background] Abdulhadi B, Abdullah M, Alaki S, Alamoudi N, Attar M. Clinical evaluation between zirconia crowns and stainless steel crowns in primary molars teeth. J Pediatr Dent. 2017;5(1):21.
- [Background] Ashima G, Sarabjot KB, Gauba K, Mittal HC. Zirconia crowns for rehabilitation of decayed primary incisors: an esthetic alternative. J Clin Pediatr Dent. 2014 Fall;39(1):18-22. doi: 10.17796/jcpd.39.1.t6725r5566u4330g. PMID 25631720
- [Background] Schweiger J, Edelhoff D, Guth JF. 3D Printing in Digital Prosthetic Dentistry: An Overview of Recent Developments in Additive Manufacturing. J Clin Med. 2021 May 7;10(9):2010. doi: 10.3390/jcm10092010. PMID 34067212